CLINICAL TRIAL: NCT01001208
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Adding Methotrexate to Etanercept in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: The Efficacy and Safety of Adding Methotrexate to Etanercept in Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Immunex Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20070559
Record Dates: First submitted 2009-10-15; First posted 2009-10-26 (Estimated); Results first posted 2013-08-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-07

CONDITIONS: Psoriasis
Keywords: Etanercept; Methotrexate; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Methotrexate; Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Etanercept Plus Methotrexate (Experimental): Participants received 50 mg etanercept twice weekly (BIW) for the first 12 weeks and then 50 mg etanercept once weekly (QW) for the second 12 weeks. Participants also received active methotrexate titrated as follows: 7.5 mg per week (3 capsules) for weeks 1 and 2, 10 mg per week (4 capsules) for weeks 3 and 4, and then up to 15 mg per week (6 capsules) or the maximum tolerated dose for the remainder of the 24-week treatment period.
  Interventions: Drug: Methotrexate; Drug: Etanercept
- Etanercept Plus Placebo (Active Comparator): Participants received 50 mg etanercept twice weekly (BIW) for the first 12 weeks and then 50 mg etanercept once weekly (QW) for the second 12 weeks. Participants also received oral placebo that was the same number of capsules per week as the methotrexate dosing regimen.
  Interventions: Drug: Etanercept; Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate — Methotrexate tablets over-encapsulated for blinding
  Arms: Etanercept Plus Methotrexate
Drug: Etanercept — 1 mL for subcutaneous injection
  Other Names: Enbrel
Drug: Placebo — Matching placebo to methotrexate capsules
  Arms: Etanercept Plus Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of adding methotrexate to etanercept compared with etanercept monotherapy as measured by the percentage of participants achieving a 75% improvement from baseline in the Psoriasis Area and Severity Index (PASI 75) at Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Is capable of understanding and giving written, voluntary informed consent before study screening
* Male or female ≥18 years of age at time of screening
* Has had stable moderate to severe plaque psoriasis for at least 6 months (eg, no morphology changes or significant flares of disease activity)
* Has involved body surface area (BSA) ≥ 10% and Psoriasis Area and Severity Index (PASI) ≥ 10 at screening and at baseline
* Is a candidate for systemic therapy or phototherapy in the opinion of the investigator
* Has a negative test for hepatitis B surface antigen and hepatitis C antibody
* Has a negative purified protein derivative test within 30 days prior to the first IP dose. Tuberculin skin tests should be considered positive when they have greater than or equal to 5 mm of induration at 48-72 hours after test is placed. Patients with a positive tuberculin skin test (if less than or equal to 14 mm of induration) are allowed if they have a history of Bacillus Calmette-Guerin vaccination with a negative Quantiferon test in the past year, no symptoms per tuberculosis worksheet, and a negative chest X ray.
* Has a negative serum pregnancy test within 28 days before initiating Investigational Product (IP) and negative urine pregnancy test at baseline for females (except those at least 3 years post menopausal or surgically sterile)
* Females are willing to use highly effective form of birth control (decided upon with the investigator) during the study and for 3 months after the end of treatment (except women at least 3 years post menopausal or surgically sterile)
* Males are willing to use highly effective form of birth control (decided upon with the investigator) during the study and for 5 months after the end of treatment (except for men who are surgically sterile or whose female partners are at least 3 years post menopausal, surgically sterile, or are using a highly effective form of birth control)
* Men with a pregnant female partner are willing to use effective methods (decided upon with the investigator) to ensure that an unborn child is not exposed to IP via semen
* Patient or designee must have the ability to inject etanercept subcutaneously

Exclusion Criteria:

Skin-disease related

* Has active guttate, erythrodermic, or pustular psoriasis at the time of the screening visit.
* Has evidence of skin conditions at the time of the screening visit (eg, eczema) that would interfere with evaluations of the effect of IP on psoriasis.

Medical conditions

* Has significant concurrent medical conditions, including:
* Type 1 diabetes
* Poorly controlled type 2 diabetes (hemoglobin A1c > 8.5)
* Symptomatic heart failure (New York Heart Association [NYHA] class II, III, or IV)
* Myocardial infarction within the last year
* Current or history of unstable angina pectoris within the last year
* Uncontrolled hypertension as defined by a resting blood pressure ≥ 160/95 mmHg prior to randomization (confirmed by a repeat assessment)
* Severe chronic pulmonary disease (eg, requiring oxygen therapy)
* No major chronic inflammatory disease or connective tissue disease other than psoriasis and/or psoriatic arthritis
* Multiple sclerosis or any other demyelinating disease
* Active malignancy, including evidence of cutaneous basal or squamous cell carcinoma or melanoma, or history of cancer (other than fully resected and surgically cured cutaneous basal cell and squamous cell carcinoma) within 5 years before the first IP dose. If malignancy occurred more than 5 years ago, documentation of disease-free state since treatment is required.
* Known immunodeficiency syndromes including human immunodeficiency virus (HIV)
* Uncontrolled, clinically significant history of renal disease
* Alcoholic hepatitis
* Any condition that, in the opinion of the investigator, might cause this study to be detrimental to the patient
* Has any active CTC grade 2 or higher infection (including chronic or localized infections) within 30 days prior to screening, at screening, or during screening period prior to first investigational product (IP) dose
* Is pregnant or breast feeding
* Has any condition that could, in the opinion of the investigator, compromise the patient's ability to give written consent and/or comply with the study procedures, such as a history of substance abuse or a psychiatric condition Methotrexate contraindications or precautions
* Has a family history of heritable liver disease (eg, hemachromatosis, Wilson's disease)
* Has a history of or evidence at screening or baseline of alcohol abuse, alcoholic liver disease, or other clinically significant liver disease
* Is unwilling or unable to limit alcohol consumption during the 24-week trial period (allowable limits are: not more than 4 drinks a week, not more than 2 drinks in a single day. 1 drink = 1 (5 oz) glass of wine = 1.5 oz liquor = 12 oz of beer or hard cider)
* Has an estimated total cumulative methotrexate exposure (by medical history) exceeding 1000 mg, unless a subsequent liver biopsy has demonstrated no grade IIIb or greater injury
* Has a history of significant methotrexate toxicity including pneumonitis or significant cytopenias

Laboratory abnormalities

* Has laboratory abnormalities at screening, including:
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > the upper limit of normal (if screen fail for abnormal AST/ALT, 1 repeat measurement is allowed)
* Serum total bilirubin ≥ 1.5 mg/dL
* Abnormal serum albumin (< 3.5 g/dL)
* Hemoglobin < 11 g/dL
* Platelet count < 125,000 /mm^3
* White blood cell count < 3,500 cells/mm^3
* Absolute neutrophil count < 1500/mm^3
* Estimated creatinine clearance < 50 mL/min (Cockroft-Gault formula, calculated value to be provided to sites)
* Any other laboratory abnormality, which, in the opinion of the investigator, will prevent the patient from completing the study or will interfere with the interpretation of the study results

Washouts and disallowed medications

* Has used any of the following therapies within 14 days of IP initiation:
* Ultraviolet light B therapy
* Topical cyclosporine or calcineurin inhibitors
* Topical vitamin A or D analog preparations
* Class III through VII topical steroids (exception: permitted on the scalp, axillae, and groin)
* Has used any of the following therapies within 28 days of IP initiation:
* Intravenous or oral calcineurin inhibitors
* Ultraviolet light A therapy
* Psoralen and ultraviolet light A therapy
* Oral retinoids
* Class I or II topical steroids
* Anthralin
* Any other systemic psoriasis therapy (eg, cyclosporine), including oral or parenteral corticosteroids
* Cyclophosphamide
* Sulfasalazine
* Has used methotrexate within 28 days of IP initiation. Patients with prior use of methotrexate must be excluded if subject discontinued because of a clinically significant adverse event (eg, severe skin reactions, methotrexate-induced lung disease, or any other adverse event that the investigator feels might cause this study to be detrimental to the patient)
* Has used biologic therapies (other than interleukin (IL)12/IL23 inhibitors or anti-timor necrosis factor (TNF) agents) within 3 months of IP initiation
* Has used an IL12/23 inhibitor within 6 months of IP initiation (eg, CNTO 1275, ABT 874)
* Has used one or more anti-TNF agents (eg, etanercept, adalimumab, infliximab) within 3 months of IP initiation. Patients with prior use of an anti-TNF agent must be excluded if the subject discontinued for lack of efficacy or a clinically significant adverse event (eg, serious infection, neurologic event, malignancy, hematologic event, or any other adverse event that the investigator feels might cause this study to be detrimental to the patient).
* Has previously used efalizumab (Raptiva®).
* Other investigational procedures are excluded.
* currently enrolled in or has not yet completed at least 30 days or 5 half-lives (if applicable; whichever is longer) since ending other investigational device or drug study(s), or is receiving other investigational agent(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 09 November 2009 through 25 June 2010
Groups:
- Etanercept + Methotrexate: Participants received 50 mg etanercept twice weekly (BIW) for the first 12 weeks and then 50 mg etanercept once weekly (QW) for the second 12 weeks. Participants also received active methotrexate titrated as follows: 7.5 mg per week (3 capsules) for weeks 1 and 2, 10 mg per week (4 capsules) for weeks 3 and 4, and then up to 15 mg per week (6 capsules) or the maximum tolerated dose for the remainder of the 24-week treatment period.
- Etanercept + Placebo: Participants received 50 mg etanercept twice weekly (BIW) for the first 12 weeks and then 50 mg etanercept once weekly (QW) for the second 12 weeks. Participants also received oral placebo that was the same number of capsules per week as the methotrexate dosing regimen.
Period: Overall Study
Arm/Group | Etanercept + Methotrexate | Etanercept + Placebo
Started | 239 | 239
Completed | 211 | 206
Not Completed | 28 | 33
Not completed — Adverse Event | 10 | 5
Not completed — Lost to Follow-up | 5 | 9
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Ineligibility Determined | 4 | 2
Not completed — Noncompliance | 4 | 7
Not completed — Disease Progression | 0 | 3
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept + Methotrexate | Etanercept + Placebo | Total
Number analyzed (Participants) | 239 | 239 | 478
Age Continuous [Mean (Standard Deviation); unit: years] | 42.99 (13.06) | 45.23 (12.79) | 44.11 (12.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 72 | 158
  Male | 153 | 167 | 320
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 10 | 9 | 19
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 4 | 10 | 14
  White | 179 | 177 | 356
  Hispanic or Latino | 42 | 39 | 81
  Japanese | 0 | 0 | 0
  Other | 1 | 3 | 4
  Aborigine | 0 | 0 | 0
Psoriasis Area and Severity Index (PASI) Score [Mean (Standard Deviation); unit: Units on a scale] — Psoriasis Area and Severity Index (PASI) Score incorporates measures of erythema, desquamation, infiltration, and affected body surface area. Involvement and severity of psoriasis was scored by physicians using a scale of 0 to 72, where 0 = no psoriasis and 72 = severe disease.
  Units on a scale | 18.24 (8.15) | 18.34 (6.62) | 18.29 (7.42)
Percent of Body Surface Area (BSA) Involved in Psoriasis [Mean (Standard Deviation); unit: Percentage of BSA] | 24.43 (15.94) | 24.23 (13.64) | 24.33 (14.82)
Body Mass Index Group [Number; unit: participants]
  <=35 kg/m^2 | 172 | 173 | 345
  >35 kg/m^2 | 67 | 66 | 133
Prior Anti-tumor Necrosis Factor (TNF) Exposure [Number; unit: participants]
  Yes | 42 | 48 | 90
  No | 197 | 191 | 388

OUTCOME MEASURES:

1. Primary Outcome: PASI 75 Response at Week 24
Description: Percentage of participants achieving at least a 75% decrease (improvement) from Baseline in the Psoriasis Area and Severity Index (PASI) at Week 24. PASI Score incorporates measures of erythema, desquamation, infiltration, and affected body surface area. Involvement and severity of psoriasis was scored by a blinded assessor using a scale of 0 to 72, where 0 = no psoriasis and 72 = severe disease.
Time Frame: Baseline and 24 Weeks
Population: Intention-to-Treat with available data; last observation carried forward (LOCF) imputation was used.
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept + Methotrexate | Etanercept + Placebo
Number analyzed (Participants) | 238 | 234
Percentage of participants | 77.3 | 60.3
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs Etanercept + Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Overall significance level for primary and secondary endpoints controlled based on a combination of sequential testing and Hommel procedures; Stratified by baseline body mass index group and prior anti-TNF exposure group

2. Secondary Outcome: PASI 50 Response at Week 24
Description: Percentage of participants achieving at least a 50% decrease (improvement) from Baseline in the Psoriasis Area and Severity Index (PASI) at Week 24. PASI Score incorporates measures of erythema, desquamation, infiltration, and affected body surface area. Involvement and severity of psoriasis was scored by a blinded assessor using a scale of 0 to 72, where 0 = no psoriasis and 72 = severe disease.
Time Frame: Baseline and 24 Weeks
Population: Intention-to-Treat with available data; last observation carried forward (LOCF) imputation was used.
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept + Methotrexate | Etanercept + Placebo
Number analyzed (Participants) | 238 | 234
Percentage of participants | 91.6 | 84.6
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs Etanercept + Placebo; Test type: Superiority or Other; p = 0.0112, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by baseline body mass index group and prior anti-TNF exposure group

3. Secondary Outcome: Static Physician Global Assessment (sPGA) Response at Week 24
Description: Percentage of participants achieving a clear (0) or almost clear (1) status on the Static Physician Global Assessment (sPGA) at Week 24. This index evaluates the physician's global assessment of the participant's psoriasis based on severity of induration, scaling, and erythema. The assessment was scored by a blinded assessor on a scale of 0 to 5, where 0 = clear, with no evidence of plaque elevation, erythema, or scale, and 5 = severe induration, erythema, and scaling.
Time Frame: Week 24
Population: Intention-to-Treat with available data; last observation carried forward (LOCF) imputation was used.
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept + Methotrexate | Etanercept + Placebo
Number analyzed (Participants) | 238 | 234
Percentage of participants | 71.8 | 54.3
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs Etanercept + Placebo; Test type: Superiority or Other; p = 0.0112, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by baseline body mass index group and prior anti-TNF exposure group

4. Secondary Outcome: PASI 50 Response at Week 12
Description: Percentage of participants achieving at least a 50% decrease (improvement) from Baseline in the Psoriasis Area and Severity Index (PASI) at Week 12. PASI Score incorporates measures of erythema, desquamation, infiltration, and affected body surface area. Involvement and severity of psoriasis was scored by a blinded assessor using a scale of 0 to 72, where 0 = no psoriasis and 72 = severe disease.
Time Frame: Baseline and 12 Weeks
Population: Intention-to-Treat with available data; last observation carried forward (LOCF) imputation was used.
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept + Methotrexate | Etanercept + Placebo
Number analyzed (Participants) | 238 | 234
Percentage of participants | 92.4 | 83.8
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs Etanercept + Placebo; Test type: Superiority or Other; p = 0.0112, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by baseline body mass index group and prior anti-TNF exposure group

5. Secondary Outcome: PASI 75 Response at Week 12
Description: Percentage of participants achieving at least a 75% decrease (i.e. improvement) from Baseline in the Psoriasis Area and Severity Index (PASI) at Week 12. PASI Score incorporates measures of erythema, desquamation, infiltration, and affected body surface area. Involvement and severity of psoriasis was scored by a blinded assessor using a scale of 0 to 72, where 0 = no psoriasis and 72 = severe disease.
Time Frame: Baseline and 12 Weeks
Population: Intention-to-Treat with available data; last observation carried forward (LOCF) imputation was used
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept + Methotrexate | Etanercept + Placebo
Number analyzed (Participants) | 238 | 234
Percentage of participants | 70.2 | 54.3
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs Etanercept + Placebo; Test type: Superiority or Other; p = 0.0112, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by baseline body mass index group and prior anti-TNF exposure group

6. Secondary Outcome: Static Physician Global Assessment (sPGA) Response at Week 12
Description: Percentage of participants achieving a clear (0) or almost clear (1) status on the Static Physician Global Assessment (sPGA) at Week 12. This index evaluates the physician's global assessment of the participant's psoriasis based on severity of induration, scaling, and erythema. The assessment was scored by a blinded assessor on a scale of 0 to 5, where 0 = clear, with no evidence of plaque elevation, erythema, or scale, and 5 = severe induration, erythema, and scaling.
Time Frame: Week 12
Population: Intention-to-Treat with available data; last observation carried forward (LOCF) imputation was used.
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept + Methotrexate | Etanercept + Placebo
Number analyzed (Participants) | 238 | 234
Percentage of participants | 65.5 | 47
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs Etanercept + Placebo; Test type: Superiority or Other; p = 0.0112, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by baseline body mass index group and prior anti-TNF exposure group

7. Secondary Outcome: PASI 90 Response at Week 12
Description: Percentage of participants achieving at least a 90% decrease (improvement) from Baseline in the Psoriasis Area and Severity Index (PASI) at Week 12. PASI Score incorporates measures of erythema, desquamation, infiltration, and affected body surface area. Involvement and severity of psoriasis was scored by a blinded assessor using a scale of 0 to 72, where 0 = no psoriasis and 72 = severe disease.
Time Frame: Baseline and 12 Weeks
Population: Intention-to-Treat with available data; last observation carried forward (LOCF) imputation was used.
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept + Methotrexate | Etanercept + Placebo
Number analyzed (Participants) | 238 | 234
Percentage of participants | 34 | 23.1
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs Etanercept + Placebo; Test type: Superiority or Other; p = 0.0348, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by baseline body mass index group and prior anti-TNF exposure group

8. Secondary Outcome: PASI 90 Response at Week 24
Description: Percentage of participants achieving at least a 90% decrese (improvement) from Baseline in the Psoriasis Area and Severity Index (PASI) at Week 24. PASI Score incorporates measures of erythema, desquamation, infiltration, and affected body surface area. Involvement and severity of psoriasis was scored by a blinded assessor using a scale of 0 to 72, where 0 = no psoriasis and 72 = severe disease.
Time Frame: Baseline and 24 Weeks
Population: Intention-to-Treat with available data; last observation carried forward (LOCF) imputation was used.
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept + Methotrexate | Etanercept + Placebo
Number analyzed (Participants) | 238 | 234
Percentage of participants | 53.8 | 34.2
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs Etanercept + Placebo; Test type: Superiority or Other; p = 0.0112, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Stratified by baseline body mass index group and prior anti-TNF exposure group

9. Secondary Outcome: Change From Baseline in the Percentage of Body Surface Area Involved With Psoriasis at Week 12
Description: A measurement of psoriasis involvement, given as the physician's assessment of the percentage of the participant's total body surface area (BSA) involved with psoriasis. The BSA numerical score was completed by a blinded assessor. A decrease from Baseline indicates improvement. Change from Baseline was calculated as Baseline score - Week 12 score; a positive change from Baseline therefore indicates improvement.
Time Frame: Baseline and 12 Weeks
Population: Intention-to-Treat with available data; last observation carried forward (LOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: Percentage of BSA
Arm/Group | Etanercept + Methotrexate | Etanercept + Placebo
Number analyzed (Participants) | 238 | 234
Percentage of BSA | 16.3 (13.7) | 15.2 (13.4)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs Etanercept + Placebo; Test type: Superiority or Other; p = 0.1995, 2-sided van Elteren test — [p-value comment as in outcome 1, analysis 1]; Stratified by baseline body mass index group and prior anti-TNF exposure group

10. Secondary Outcome: Change Form Baseline in Percentage of Body Surface Area Involved With Psoriasis at Week 24
Description: A measurement of psoriasis involvement, given as the physician's assessment of the percentage of the participant's total body surface area (BSA) involved with psoriasis. The BSA numerical score was completed by a blinded assessor. A decrease from Baseline indicates improvement. Change from Baseline was calculated as Baseline score - Week 24 score; a positive change from Baseline therefore indicates improvement.
Time Frame: Baseline and 24 Weeks
Population: Intention-to-Treat with available data; last observation carried forward (LOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: Percentage of BSA
Arm/Group | Etanercept + Methotrexate | Etanercept + Placebo
Number analyzed (Participants) | 238 | 234
Percentage of BSA | 19.5 (15.2) | 17.8 (14.0)
Statistical Analysis 1: Comparison: Etanercept + Methotrexate vs Etanercept + Placebo; Test type: Superiority or Other; p = 0.1995, 2-sided van Elteren test — [p-value comment as in outcome 1, analysis 1]; Stratified by baseline body mass index group and prior anti-TNF exposure group

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Etanercept + Placebo | Etanercept + Methotrexate
Serious Adverse Events (participants affected / at risk) | 3/239 | 2/239
Other Adverse Events (participants affected / at risk) | 58/239 | 67/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept + Placebo (N=239) | Etanercept + Methotrexate (N=239)
Myocardial Infarction (Cardiac disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Pneumonia Bacterial (Infections and infestations) | 0 | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept + Placebo (N=239) | Etanercept + Methotrexate (N=239)
Nausea (Gastrointestinal disorders) | 7 | 13
Nasopharyngitis (Infections and infestations) | 26 | 23
Upper Respiratory Tract Infection (Infections and infestations) | 12 | 20
Headache (Nervous system disorders) | 22 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial resul